CLINICAL TRIAL: NCT01728935
Title: Serologic and Virologic Outcomes of Tenofovir in Asian Chronic Hepatitis B Patients With Prior Nucleoside Analogue Exposure
Brief Title: Tenofovir in Asian Chronic Hepatitis B Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDF-HKU; UW 11-241 (Other: Institutional Review Board The University of Hong Kong / Hospital Authority Hong Kong West Cluster)
Record Dates: First submitted 2012-11-08; First posted 2012-11-20 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis B
Keywords: HBV; Tenofovir; HBV DNA; HBsAg; Resistance
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

ARMS (1):
- Tenofovir disoproxil (Other): Tenofovir disoproxil 300mg daily
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil — Tenofovir disoproxil 300mg daily
  Other Names: Viread

SUMMARY:
Tenofovir (TDF) has been demonstrated to have potency antiviral against the hepatitis B virus (HBV) in various multiple-centre trials, with no cases of resistance encountered. However, its efficacy and resistance profile in the Asian population, which constitute the majority of chronic hepatitis B (CHB) patients, is unknown. Compared to other nucleoside analogues, TDF has been associated with relatively high rates of hepatitis B surface antigen (HBsAg) seroclearance. It would be interested to see if this could be reproduced. The investigators plan to report the serologic and virologic results of our 140 nucleoside analogue-experienced patients who were commenced on TDF.

DETAILED DESCRIPTION:
Recent multi-center trials have shown tenofovir disoprovil fumarate (TDF) demonstrating potent antiviral efficacy in both nucleoside-naive and -experienced chronic hepatitis B (CHB) patients. At present, there has been no identifiable amino acid substitutions associated with resistance to TDF.

Since TDF and adefovir (ADV), another licensed drug for CHB, belong to same molecular group, acyclic phosphonate, there had been various studies investigating the efficacy of TDF in ADV-resistant patients. The efficacy of tenofovir in this group of patients is conflicting. While several studies have shown TDF achieving similar viral suppression when compared to CHB patients without ADV-resistance , another study found that patients with the signature ADV mutations of rtA181V/T and /or rtN236T responded suboptimally to TDF. For all published studies, the number of patients with documented genotypic resistance to adefovir is actually small (n = 17-40), and therefore, further studies in this area are required.

Another interesting point to note was the relatively high rate of hepatitis B surface antigen (HBsAg) seroclearance found in patients taking TDF. The cumulative rate of HBsAg seroclearance up in hepatitis B e antigen (HBeAg)-positive was 10% after 4 years . However, the same study did not find any HBeAg-negative patients achieving HBsAg seroclearance. In addition, studies on TDF were mainly performed in Caucasian patients, the majority being genotypes A and D. A preliminary study performed in Asian patients, predominantly genotypes B and C, did not discover any cases of HBsAg seroclearance . Given the majority of the CHB population is found in Asia, further studies are needed to clarify if HBsAg seroclearance by nucleoside / nucleotide analogues is potentially achievable using TDF.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg-positivity for at least 6 months at presentation
2. Commenced on tenofovir for chronic hepatitis B
3. Exposure to other nucleoside analogues before starting TDF

Exclusion Criteria:

1. Concomitant liver diseases including chronic hepatitis C and/ or D infection, Wilson's disease, autoimmune hepatitis, primary biliary cirrhosis and primary sclerosing cholangitis.
2. Significant alcohol intake (> 20 grams per day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Serum HBV DNA levels | 3 Years

SECONDARY OUTCOMES:
Resistance Profile | 3 Years
  Performed using a Line Probe Assay (LiPA)
HBsAg levels | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Man-Fung Yuen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong